CLINICAL TRIAL: NCT06709677
Title: Prevalence of Musculoskeletal Disorders Among Egyptian Students in the Faculty of Applied Arts
Brief Title: Prevalence of Musculoskeletal Disorders
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Osama Abdelaziz, physical therapy practitioner, Cairo University
Other Study IDs: P.T.REC/012/005019
Record Dates: First submitted 2024-11-26; First posted 2024-11-29 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Musculoskeletal Disorders; Among Egyptian Students in the Faculty of Applied Arts
Keywords: Prevalence; Musculoskeletal Disorders; Egyptian Students; Faculty of Applied Arts
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Behavioral: Arabic version of The Nordic Musculoskeletal Questionnaire (NMQ) is a standardized questionnaire used to assess musculoskeletal symptoms and disorders in the workplace — The Nordic Musculoskeletal Questionnaire (NMQ) is a standardized questionnaire used to assess musculoskeletal symptoms and disorders in the workplace. It is commonly used in occupational health and ergonomic assessments to gather information about the prevalence and severity of musculoskeletal issues such as pain, discomfort, and limitations in movement. The NMQ typically includes questions about specific body regions (e.g. neck, shoulders, back, wrists) and asks individuals to report any symptoms they may be experiencing in those areas. This information can help identify potential risk factors for musculoskeletal disorders and guide interventions to prevent or manage these conditions in the workplace (Namnik et al., 2016).
  • Section 1: a general questionnaire of 40 forced-choice items identifying areas of the body causing musculoskeletal problems. Completion is aided by a body map to indicate nine symptom sites being neck, shoulders, upper back, elbows, low back, wrist/hands, hips/thi

SUMMARY:
This observational cross-sectional study aims to determine the prevalence of musculoskeletal disorders (MSDs) among Egyptian students in the Faculty of Applied Arts. Using the Arabic version of the extended Nordic Musculoskeletal Questionnaire (NMQ-E), the study will assess the prevalence, distribution, and associated factors of musculoskeletal symptoms over the last 12 months and 7 days. A sample of 250 participants, aged 20-22 years and of both genders, will be recruited. Exclusion criteria include obesity, pregnancy, history of neuropathy, unstable medical conditions, or trauma-related musculoskeletal problems. The results will provide insights into MSD prevalence and help guide interventions for this population.

DETAILED DESCRIPTION:
Study Title: Prevalence of Musculoskeletal Disorders Among Egyptian Students in the Faculty of Applied Arts

Study Design:

This is an observational, cross-sectional study aimed at investigating the prevalence of musculoskeletal disorders (MSDs) and associated risk factors among Egyptian students enrolled in the Faculty of Applied Arts during their last three academic years. The study will collect demographic data (age, gender) and assess musculoskeletal symptoms using the Nordic Musculoskeletal Questionnaire (NMQ-E).

Study Population:

The target population includes approximately 9,600 students from the Faculty of Applied Arts in Egypt. A sample of 250 participants will be recruited based on eligibility criteria.

Inclusion Criteria:

Egyptian students from the Faculty of Applied Arts. Age range: 20-22 years. Both genders included.

Exclusion Criteria:

Obesity. Pregnancy. History of neuropathy or other neurological disorders such as lumbar plexopathy, spinal stenosis, and nerve root compression.

Unstable medical conditions. History of central nervous system malignancy (primary or metastatic). Musculoskeletal problems due to trauma or previous surgery.

Sample Size Calculation:

The sample size was determined using a sample size calculator with a confidence interval of 95% and α level of 0.05. From a population of 9,600, a minimum of 250 participants was required to achieve statistical power.

Instrumentations:

The Arabic version of the extended Nordic Musculoskeletal Questionnaire (NMQ-E) will be utilized. The NMQ is a validated tool for assessing musculoskeletal symptoms, including pain prevalence and anatomical distribution.

Key Sections of NMQ-E:

Section 1: 40 forced-choice items identifying musculoskeletal problem areas, supported by a body map. Symptoms over the last 12 months and the past 7 days will be evaluated.

Section 2: Additional questions on neck, shoulders, and lower back, covering symptom duration, functional impact, professional assessments, and recent musculoskeletal problems.

Procedure:

Participants will be recruited from the Faculty of Applied Arts and asked to complete the NMQ-E online or in person. Data on musculoskeletal symptoms and ergonomic practices will be collected over a specific timeframe.

Validity and Reliability of NMQ-E:

Validity:

Content validity is supported by expert review and alignment with established measures of musculoskeletal health.

Criterion validity demonstrated strong correlations between NMQ responses and clinical assessments (sensitivity: 66-92%; specificity: 71-88%).

Reliability:

High test-retest reliability observed in various populations. Internal consistency confirmed via Cronbach's alpha.

Data Analysis and Statistical Design:

The collected data will be analyzed using statistical software, employing:

Descriptive statistics (mean, standard deviation, percentages). Statistical significance set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. 250 Egyptian students from different Faculties of Applied Art.
2. Age (20-22) years old
3. both genders will be included.

Exclusion Criteria:

1. Obesity.
2. Pregnancy.
3. Patients who had history of any other neuropathy.
4. Unstable medical condition.
5. Other neurological disorders causing pain as lumbar plexopathy, spinal stenosis, and spinal nerve root compression.
6. History of central nervous system primary or metastatic malignancy
7. student having any musculoskeletal problems due to other causes as accidents or a previous operation.

Ages: 20 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: students enrolled in the Faculty of Applied Art at a university in Egypt
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-01-05 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
musculoskeletal symptoms | one month
  information on musculoskeletal symptoms experienced by participants,